CLINICAL TRIAL: NCT04042987
Title: Assessing Malnutrition Prevalence and Impact of a Nutrition-Focused Quality Improvement Program (QIP) Among Community-Dwelling Malnourished Colombian Patients Receiving Care in an Ambulatory Health Clinic
Brief Title: Nutrition-Focused Quality Improvement Program (QIP) Among Community Dwelling Malnourished Patients
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: Hospital Universitario San Ignacio, Aging Institute, Pontificia Universidad Javeriana (Unknown)
Responsible Party: Sponsor
Other Study IDs: HA38
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical Control Group: Retrospective chart review
- Prospective QIP Group: Participants that meet eligibility criteria will be prospectively enrolled into QIP including malnutrition screening, nutrition consultation, expedited provision of oral nutritional supplementation (ONS) and encouragement of ONS consumption.

SUMMARY:
This study aims to assess the malnutrition prevalence of Colombian community-dwelling adults and evaluate the feasibility of a nutrition-focused QIP implemented in a Colombian ambulatory care facility on healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient is screened as being malnourished or at risk for malnutrition
* Patient can consumer beverages and food orally
* Patients have a life expectancy of equal or greater than 90 days
* Patient is literate and willing to voluntarily sign and date an Informed Consent Form (ICF) after it is explained

Exclusion Criteria:

* Patient is pregnant
* Patient is intubated, receiving tube feeding or parenteral nutrition
* Patient has severe dementia, delirium or history of significant psychiatric disorder and no dedicated caregiver who could assure their compliance with QIP study requirements and help with the completion of QIP study materials
* Any other disorder that may interfere with QIP product consumption or compliance with QIP protocol procedures
* Patient has an allergy or intolerance to any of the ONS ingredients
* Patients does not want to participate or sign ICF
* Patient is bedridden or confined in a wheelchair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sites will recruit patients for QIP group at discharge from hospital (after 3 months) or in ambulatory care facility.
Sampling Method: Non-Probability Sample
Enrollment: 1325 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of Malnutrition | Change from Baseline to Week 10 post-QIP enrollment
  Measured by the Mini Nutritional Assessment (MNA®) a maximum 30 point scale resulting in a single Malnutrition Indicator Score where lower number indicates malnutrition

SECONDARY OUTCOMES:
Healthcare Resource Utilization | 10-weeks follow-up period post enrollment from ambulatory care facility
  Chart Review

OTHER OUTCOMES:
Body mass index (BMI) | Baseline and Week 10 post-QIP enrollment
  BMI calculated Weight (kg)/Height (m)2
Calf Circumference (CC) | Baseline and Week 10 post-QIP enrollment
  Measurement at largest circumference of calf
Short Physical Performance Battery (SPPB) | Baseline and Week 10 post-QIP enrollment
  Timed assessments of balance, gait speed and chair standing; Scaled in the negative direction
Hand Grip | Baseline and Week 10 post-QIP enrollment
  Participant assessed with hand dynamometers
Quality of Life EuroQOL EQ-5D | Baseline and Week 10 post-QIP
  Subject rated health state of 5 dimensions. Each dimension has 5-levels scaled in negative direction resulting in an overall 5-digit number describing the health state; EQ VAS Score 0-100 points scaled in positive direction
Nutritional Supplement Consumption | Baseline and Week 10 post-QIP
  Participant reported

CONTACTS AND LOCATIONS:
Overall Officials: Suela Sulo, PhD, MSc, Study Chair — Abbott Nutrition
Locations (1):
- Geriatric Unit. Hospital Universitario San Ignacio, Aging Institute, Pontificia Universidad Javeriana, Bogotá, Colombia

REFERENCES:
- [Derived] Gomez G, Botero-Rodriguez F, Misas JD, Garcia-Cifuentes E, Sulo S, Brunton C, Venegas-Sanabria LC, Gracia DA, Cano Gutierrez CA. A nutritionally focused program for community-living older adults resulted in improved health and well-being. Clin Nutr. 2022 Jul;41(7):1549-1556. doi: 10.1016/j.clnu.2022.05.003. Epub 2022 May 13. PMID 35667271
- [Derived] Chavarro-Carvajal DA, Ayala AM, Venegas-Sanabria LC, Gomez G, Sulo S, Misas JD, Cano-Gutierrez C. Use of a nutrition-focused quality improvement program for community-living older adults at malnutrition risk is associated with better nutritional outcomes. Clin Nutr ESPEN. 2022 Apr;48:291-297. doi: 10.1016/j.clnesp.2022.01.032. Epub 2022 Feb 2. PMID 35331504